CLINICAL TRIAL: NCT04985994
Title: Exploring the Role of Microbiome in Susceptibility, Treatment Response and Outcome Among Tuberculosis Patients; a Prospective Cohort Study
Brief Title: Potential Role of Microbiome in Tuberculosis
Acronym: Micro-STOP
Status: Completed | Type: Observational
Sponsor: Khyber Medical University Peshawar (Other)
Collaborators: University of Reading (Other); TB Control Program Khyber Pakhtunkhwa (Unknown)
Responsible Party: Principal Investigator, Muhammad Shahzad, Associate Professor, Khyber Medical University Peshawar
Other Study IDs: DIR/KMU-EB/PR/000858; 10289/KPK/NRPU/R&D/HEC/2019 (Other Grant/Funding Number: Higher Education Commission Pakistan)
Record Dates: First submitted 2021-07-22; First posted 2021-08-02 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Pulmonary TB; Microbiome; Immunity; Nutrition; Treatment response; Treatment Outcome; Gut microbiome; Oral Microbiome; Inflammation; Dietary intake
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool, Whole Blood, Salivary rinse
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tuberculosis Patients: 1. Diagnosed with pulmonary TB after detailed history collection, clinical examination, and laboratory assessment (sputum culture positive).
  2. Aged 18 years or above.
  3. Willing to participate in the study.
- Healthy Volunteers: 1. Healthy subjects with no symptoms or history of pulmonary TB
  2. Negative sputum culture
  3. Matched for sex and age (±5 years) with the TB patient group.

SUMMARY:
Tuberculosis (TB), caused by Mycobacterium tuberculosis (Mtb), is a deadly infectious disease and major global public health problem. Recent evidence from animal studies suggests that the microbiome plays a role in TB pathogenesis and immune response. However, until now, no similar study has been performed in humans and thus any influence of the microbiota on TB or vice versa remains unknown.

DETAILED DESCRIPTION:
Tuberculosis is among one of the most difficult to treat infections that require multidrug therapy for prolonged periods, in most cases 6-9 months. Treatment failure is still common and frequently observed (even where adherence to antibiotic therapy is maintained) in 15% of drug-susceptible infections and 31% for drug-resistant cases. Although poor patient compliance and the emergence of drug-resistant Mtb strains are generally implicated as a major cause of TB treatment failure, other factors such as the role of the microbiome in TB pathogenesis and reactivation are poorly considered.

The human microbiome is a consortium/collection of all microorganisms (bacteria, archaea, viruses, and fungi) colonizing different habitats in the human body such as skin, gut, and mucosal surfaces and living in a commensal relationship with each other. Emerging evidence suggests a crucial role of the microbiome in hosts physiology, nutritional status, and development of the functional immune system. Microbial dysbiosis is the change in microbial composition or functional potential that has been implicated both in infectious diseases status as well as the development of non-communicable disease in hosts ranging from immune mediated diseases to intergenerational obesity and even cancers. Microbial dysbiosis at different body sites has also been reported in TB-associated comorbidities such as diabetes mellitus and malnutrition. However, to date, the role of the microbiome and microbial dysbiosis is not clear in the context of TB infections in humans.

Therefore, this study aims to dissect the relationship between the microbiomes and its interaction with the immune system during TB infection, and anti-tuberculosis therapy in humans.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with TB after detailed history collection, clinical examination and laboratory assessment (sputum culture positive).
2. Aged 18 - 65 years.
3. Willing to participate in the study.
4. Healthy controls are those who are free of TB symptoms, healthy on physical examination and with a negative sputum culture result.

Exclusion Criteria:

1. Already on anti-TB treatment or previously treated for TB.
2. Severely anemic (Hb < 10g/dL).
3. Having diarrhea or other major gastrointestinal disorders.
4. Using or have used aminoglycoside or quinolones antibiotics in the past one month.
5. Using a medically prescribed diet or nutrition supplement.
6. Pregnant or lactating women.
7. Patients with liver or renal dysfunction, or having any other chronic disease condition.
8. Multidrug resistance TB patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be conducted primarily in three district levels (Peshawar, Mardan and Swat) TB diagnostic and treatment centers of Khyber Pakhtunkhwa province of Pakistan. These centers have been selected based on the highest TB prevalence in the year 2020
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2021-08-22 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Gut microbiome diversity and functional potential | 2 Years
  To explore the effect of TB infection and anti-tuberculosis therapy on gut microbiome diversity, functional potential and immune response in newly diagnosed TB patients from Pakistan.

SECONDARY OUTCOMES:
Baseline Gut microbiome | 1 year
  To determine gut microbiome diversity and functional potential at baseline and compare with healthy controls
Baseline Oral microbiome | 1 year
  To determine oral microbiome diversity and functional potential at baseline and compare with healthy controls
Gut microbiome and associated factors | 1 year
  3. To assess the relationship between gut microbiome and socio-demographic characteristics and dietary intake in TB patients at baseline, before the start of anti-tuberculosis treatment.
Microbial dysbiosis | Two years
  To describe the occurrence of gut microbial dysbiosis and its association with adverse reaction and treatment failure in TB patients.
Microbial signatures | 2 years
  5. To identify specific oral and gut enterotypes associated with adverse reaction and unfavorable treatment outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Shahzad, Principal Investigator — Khyber Medical University
Locations (2):
- Pakistan (2):
  - DTO Peshawar, Peshawar, Khyber Pakhtunkhwa
  - Khyber Medical University, Peshawar, Khyber Pakhtunkhwa

IPD SHARING:
Plan to Share IPD: Yes
Access to the trial IPD can be requested by qualified researchers with research or academic interests in Tuberculosis or Microbiome research. The individual researchers will be required to send an email to the principal investigator describing the need and rationale for IPD. However, the access will be provided only after the proposal and statistical analysis plan is reviewed by the principal investigator and ORIC office of Khyber Medical University. The party requesting the access will also be required to sign Data Sharing agreement and or Material transfer agreement. Before sharing, the principal investigator will make sure that the samples and data are coded and all the personal information are removed.
Supporting Information: Study Protocol, SAP
Time Frame: Within one year after the data is published
Access Criteria: The information request should be send directly to the principal investigator by email.
URL: https://kmu.edu.pk

REFERENCES:
- [Derived] Shahzad M, Andrews SC, Ul-Haq Z. Exploring the role of Microbiome in Susceptibility, Treatment Response and Outcome among Tuberculosis Patients from Pakistan: study protocol for a prospective cohort study (Micro-STOP). BMJ Open. 2022 Jun 7;12(6):e058463. doi: 10.1136/bmjopen-2021-058463. PMID 35672071
- Available data/document: Study Protocol — https://bmjopen.bmj.com/content/12/6/e058463.full — Complete study protocol has been published and can be accessed through the URL given above.